CLINICAL TRIAL: NCT00599859
Title: Differential Biologic Impact of Lactose Consumption in Lactase Persistent and Non-persistent Populations: Evaluation of Microflora and Insulin/Glycemic Response
Brief Title: Effects of Lactose on Fecal Microflora
Acronym: ELM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Collaborators: Danone Institute International (Other)
Responsible Party: Andrew Szilagyi MD, SMBD Jewish General Hospital , McGill university
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GIA-05-01; Danone Institute Mtl, Canada
Record Dates: First submitted 2008-01-10; First posted 2008-01-24 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Lactose Intolerance
Keywords: lactase; lactose; microflora
MeSH Terms: conditions — Lactose Intolerance | interventions — Lactose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants in arm 1 are grouped as lactose digesters based on genetic analysis and breath hydrogen results. In discrepant cases the genetic status is accepted. Arm 1 is initially withdrawn from dairy foods(lactose) and then asked to consume lactose 50g in divided doses mixed in water for 2 weeks.
  Interventions: Dietary Supplement: lactose
- 2 (Active Comparator): Arm 2 are lactose maldigesters: 2 interventions are a. withdrawal from lactose for 2 weeks and b. consumption of 50g lactose in divided doses mixed in water for a 2 week period.
  Interventions: Dietary Supplement: lactose

INTERVENTIONS:
Dietary Supplement: lactose — consumption of 50g lactose/day in 2 divided doses mixed in water.
  Arms: 1
Dietary Supplement: lactose — consumption of lactose 50g/day in 2 divided doses mixed in water
  Arms: 2

SUMMARY:
The genetics of lactase divides the population into 2 phenotypes: Those who can(LP) and those who cannot(LNP)digest lactose. This division may help modify disease risks according to geographic population distribution. At least some of the putative mechanism of risk modification may relate to an effect of undigested lactose on lower intestinal bacteria. The effect may provide for support of beneficial microbes. The amount of lactose reaching the colon is made easier in LNP than LP subjects who have to consume larger amounts to have meaningful spillover into the lower bowel.The current study examines whether there are quantifiable qualitative fecal bacterial differences to a standard intake of lactose(milk sugar)between these 2 different phenotypic populations. Finding of differences would lend support to the notion that for some diseases LP and LNP subjects face different risks even in an area of uniform disease risk if they consume lactose (found in dairy foods).

The primary end point is comparison of 4 groups of specific bacteria between LP and LNP participants before and after 2 weeks of lactose(in powder form mixed in water) consumption. Classification is based on genetic analysis and secondarily on breath hydrogen results. Results are compared within groups.

The secondary outcome is comparison of 4 groups of bacteria between LP and LNP subjects against each group of stool samples obtained on the first visit. Results are obtained between groups.

Additional information and other secondary outcomes are to evaluate any relationship between diet intake and the 4 groups of bacteria on the first visit

Another outcome will be to compare within groups any effect of lactose consumption on insulin and glucose levels within the 2 groups.

DETAILED DESCRIPTION:
Healthy volunteers between the ages of 18 and 49 are recruited.

1. Each participant fills a lactose targetting diet questionnaire(3 day recall).
2. A 50g lactose challenge tets is administered,breath hydrogen and symptoms are recorded for 4.5hrs.
3. Blood is drawn for analysis of lactase genetic status.
4. A stool sample is collected(10-15g)and analysed fo total anaerobes, enterococci, bifidobacteria and lactobacilli.
5. All subjects are withdrawn from dairy foods(calcium replacement suggested in diet) for 2 weeks and are aked to return to repeat parts 2 and 4.
6. A voluntary segment has glucose and insulin measured for 4 hrs via an indwelling venous catheter.
7. Subjects are asked to consume 50g lactose in divided doses for 2 further weeks
8. At the end they return and repeat sections 2 and 4 for the third time.
9. Participants who volunteered to have glucose and insulin measured repeat this segment of the study as well.

ELIGIBILITY:
Inclusion Criteria:

* 18-49 yr old male or female.
* Healthy except may take chronic thyroid or hypertension medication.

Exclusion Criteria:

* Pregnancy
* Antibiotics in last 6 weeks
* Any active illness.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2006-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
bacterial differences within the 2 groups between the 2 weeks of lactose ingestion | 2 weeks

SECONDARY OUTCOMES:
bacterial differences between the 2 groups on comparison of first stool sample | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Szilagyi, MD, Principal Investigator — SMBD Jewish General Hospital
Locations (1):
- Sir Mortimer B Davis General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Szilagyi A, Nathwani U, Vinokuroff C, Correa JA, Shrier I. The effect of lactose maldigestion on the relationship between dairy food intake and colorectal cancer: a systematic review. Nutr Cancer. 2006;55(2):141-50. doi: 10.1207/s15327914nc5502_4. PMID 17044768
- [Background] Szilagyi A, Nathwani U, Vinokuroff C, Correa JA, Shrier I. Evaluation of relationships among national colorectal cancer mortality rates, genetic lactase non-persistence status, and per capita yearly milk and milk product consumption. Nutr Cancer. 2006;55(2):151-6. doi: 10.1207/s15327914nc5502_5. PMID 17044769